CLINICAL TRIAL: NCT06232070
Title: Real World Evaluation of Lunit INSIGHT MMG Technology in a Population of Women With Breast Symptoms Referred to a "One-stop" Breast Clinic
Brief Title: Real World Evaluation of Lunit INSIGHT MMG Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lunit Inc. (Industry)
Collaborators: King's College London (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Lunit INSIGHT protocol
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Standard Pathway Arm: All participating patients will have their mammograms reported using the standard of care. The mammograms randomised to the Standard Pathway arm will be reported using the current standard of care, which involves two human readers; The readers will be blind to Lunit INSIGHT MMG report
- Lunit Assisted Arm: All participating patients will have their mammograms reported using the standard of care. Those randomised to the Lunit assisted arm will also undergo double reader process , ensuring the current standard of clinical care is provided. In addition to that, the Lunit INSIGHT MMG report will also be available to the readers. Within this arm, each reader will be presented with a Likert scale to rank their level of agreement with the Lunit INSIGHT MMG report
  Interventions: Device: Lunit INSIGHT MMG

INTERVENTIONS:
Device: Lunit INSIGHT MMG — In the Lunit Assisted arm, the radiographers will also be seeing the Lunit INSIGHT MMG reports while reading the mammograms. The standard of care will be followed in all the cases
  Groups: Lunit Assisted Arm

SUMMARY:
This study is a single-centre prospective observational cohort study designed to assess and compare the sensitivity and specificity of a Lunit INSIGHT MMG assisted human reading to the standard care double human reading process within mammography review at a "one-stop" breast clinic (non-inferiority study).

The current imaging reporting process is a sequential double read of mammography and ultrasound (if available) images, by consultant radiologists or radiographers. The first reader produces a report which is then sent to the second reader who reviews it. If the second reader agrees with the first, this is reflected in the second reader's report which translates into a decision for further action; in the event of disagreement, a third reader arbitrates and produces the final report.

In the past, breast clinics have had to resort to single reader reporting due to staff shortages and high demand. This results in delays to any further assessments that may be required. It is worth noting however that despite difficulties in meeting the target, the current clinical pathway has proven to be cost effective.

The Lunit INSIGHT MMG tool could generate benefits and potential efficiencies if it were introduced to the clinical service as an assistant reader within the mammography reporting process, by replacing one of the two human readers in the current standard of care. Before this can be assessed however, its non-inferiority in combination with a human reader in comparison to standard of care (double human reading) must first be established. This study will aim to address this issue in the first instance, maintaining standard of care for all patients seen within the 2 week wait pathway, by introducing the use of Lunit INSIGHT MMG into one of two arms within this prospective, observational parallel cohort study.

DETAILED DESCRIPTION:
The study has three main objectives, which will be met through separate sub-studies and analyses.

First, it will investigate and compare the performance of the Lunit INSIGHT MMG tool in combination with a human reader, against the current standard of care (two human readers). Quantitative data will be collected from a prospective, observational cohort study which will take place during routine clinical care at the participating site in parallel to standard care. The main aims will be:

1. To assess and compare the sensitivity and specificity of Lunit INSIGHT MMG combined with a single human reader for non-inferiority compared to double human reading
2. To assess and compare the rate of escalation to arbitration (following non-agreement) for non-inferiority of Lunit INSIGHT MMG combined with a single human reader against double human reading
3. To assess clinician reported agreement with the Lunit INSIGHT MMG report
4. To address any differences in performance characteristics as a function of patient age 6 To assess how Lunit score relates to tumour grade on biopsy

Second, the acceptability and perceptions surrounding the AI will be investigated using qualitative data obtained from patient and workforce interviews and questionnaires from the latter. The main aims will be to assess the acceptability of the Lunit INSIGHT MMG tool to patients and the workforce and explore patient and workforce perceptions surrounding it and its implementation in clinical pathways.

Third, a health economic evaluation will be carried out in a cost effectiveness analysis to assess the value of introducing the Lunit INSIGHT MMG tool at a "one-stop" breast clinic. The main aims will be two. The implementation costs of the Lunit Insight MMG tool and costs of a scan read by it, in combination with a human reader, will be compared against the cost of double human readings based on standard practices. In addition, a valuation of outcomes will also be undertaken following the lifetime of the cohort with the use of the Lunit INSIGHT MMG tool compared with standard of care.

ELIGIBILITY:
Inclusion Criteria:

Non-Inferiority Study

* Women 18 years of age or older.
* Referred to a "one-stop" breast clinic following GP appointment for breast symptoms.

Patient and workforce qualitative studies Patients: as above. Workforce: Clinical staff and other key stakeholders involved in the implementation of Lunit INSIGHT MMG both male and female

• Able to undergo mammography.

Exclusion Criteria:

Non-Inferiority Study

* Men will not be included in this study.
* Women who are not able to tolerate a mammogram or are unable to have one due to physical difficulties in engagement with the technology caused by immobility or being wheelchair bound.

Patient and workforce qualitative studies Patients: as above. Workforce: Has no connection to Lunit INSIGHT MMG implementation irrespective of being male or female

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The symptomatic breast population will be recruited from the breast service 2 week pathway referred to a 'one-stop' breast clinic
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and cost effectiveness of Lunit INSIGHT MMG | Jan-Nov 2024
  To assess and compare the sensitivity and specificity (further follow up or not) of Lunit INSIGHT MMG combined with a single human reader for non-inferiority against double human reading
Acceptability of Lunit INSIGHT MMG to patients and NHS workforce | Jan-Nov 2024
  To assess the acceptability of Lunit INSIGHT MMG to patients and NHS workforce. This will be done through a patient and workforce qualitative study involving in-depth interviews and questionnaires
Cost Effectiveness of introducing Lunit INSIGHT MMG | Jan-Nov 2024
  To assess the cost effectiveness of introducing Lunit INSIGHT MMG at the 'one-stop' breast clinic

SECONDARY OUTCOMES:
Sensitivity and specificity of the Lunit INSIGHT MMG assisted single Human reading compared to double human reading | Jan-Nov 2024
  The sensitivity and specificity of the Lunit INSIGHT MMG assisted single human reading will be compared to double human reading through ROC curve comparison
Number and proportion of non-agreement/arbitrations in the Lunit INSIGHT MMG assisted arm vs the Standard of care pathway arm | Jan-Nov 2024
  Chi squared and Wilson tests on the number and proportion of non-agreement/arbitration in the Lunit INSIGHT MMG assisted arm vs the Standard of Care pathway arm
Correlation between the Lunit INSIGHT MMG abnormality score and the level of confidence of human reader 1 in the Lunit result | Jan-Nov 2024
  Correlation between Lunit INSIGHT MMG abnormality score (percentage continuous) and the level of confidence of human reader 1 in the Lunit result as measured by Likert scale
Correlation of reader level of concern score | Jan-Nov 2024
  Correlation of reader level of concern score (categorical ordinal) with Lunit INSIGHT MMG abnormality score (percentage continuous). This can be done using tests Kendall's tau or Somers' D if the abnormality percentage are converted to categorical scores
Investigation of performance of the Lunit assisted arm in sub-categories of patients | Jan-Nov 2024
  Investigation of performance of the Lunit assisted arm in sub-categories of patients for different ages, breast density, BMI, smoking status and family history using ANOVA or Kruskal-Wallis tests
Comparison of time to final report between the two arms | Jan-Nov 2024
  Comparison of time to final report between the two arms with T-test and Mann-Whitney test.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Sharma, Principal Investigator — The Leeds Teaching Hospital NHS Trust
Locations (1):
- The Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient identifiable data will be shared outside of the direct care team for the main study. The qualitative interview data will only be available to the King's College Research team which also be anonymized after transcription.